CLINICAL TRIAL: NCT02034604
Title: Efficacy and Safety of Naftopidil in Patient With Neurogenic Lower Urinary Tract Dysfunction Not Caused by Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, KYU-SUNG LEE, professor,MD,PhD, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-02-043
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Neurogenic Lower Urinary Tract Dysfunction
Keywords: Naftopidil; safety
MeSH Terms: interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naftopidil Group (Experimental): Naftopidil medication patients
  Interventions: Drug: Naftofidil
- Tamsulosin Goup (Active Comparator): Tamsulosin medication patients
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: Naftofidil
  Arms: Naftopidil Group
Drug: Tamsulosin
  Arms: Tamsulosin Goup

SUMMARY:
This study is designed to evaluate efficacy and safety of naftopidil in patient with neurogenic lower urinary tract dysfunction not caused by benign prostatic hyperplasia.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 20 years old and above (upper limit of age: 80 years old)
2. patients diagnosed as neurogenic bladder due to cerebrovascular accident, parkinson disease, spinal cord lesion, diabetic neuropathy etc)
3. a+b

   1. IPSS ≥ 12 and QoL ≥ 3
   2. Maximum Flow Rate <15 mL/s (Voiding volume) ≥ 120mL)
4. Ability and willingness to correctly complete the micturition diary and questionnaire
5. Capable of understanding and having signed the informed consent form after full discussion of the research nature of the treatment and its risks and benefits

Exclusion Criteria:

1. In male aged 50 years old and above, bladder outlet obstruction (Bladder Outlet Obstruction Index(BOOI) ≥40)
2. In female, Pelvic Organ Prolapse ICS stage; POP-Q stage ≥ 2
3. In female, the history of anti-incontinence operation.
4. Patients with cancer of any type including cancer of the prostate or bladder
5. Patients with urethral stricture or bladder neck contracture

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2013-12; Primary Completion 2016-12 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Changes in patients' symptom questionnaires | from baseline to 8 weeks of treatment
  international prostate symptom score (IPSS) change, except QOL domain scores

SECONDARY OUTCOMES:
Changes in uroflow parameters | from baseline to 8 weeks of treatment
  maximal flow rate, mean flow rate, voided volume and Changes in uroflowmetry parameters : maximal flow rate,mean flow rate, voided volume and PVR
Change in proportion of patients showed an improvement in IPSS total scores of more than 25%. | from baseline to 8 weeks of treatment
Benefit, Satisfaction, and Willingness to Continue (BSW) questions | 8 weeks after treatment
Score of global response assessment for Korean, GRA-K | 8 weeks after treatment
Treatment satisfaction question, TSQ | 8 weeks after treatment
safety evaluation : incidence and severity of adverse events | up to 8 weeks
change in each domain scores of IPSS | up to 8 weeks
change in number of urinary frequency, nocturia | up to 8weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea